CLINICAL TRIAL: NCT02282462
Title: A Randomized Comparison of Active Suction vs. Passive Chest Tube Drainage and Regulated and Unregulated Pleural Pressure After Anatomic Lung Resection
Brief Title: Study of Postoperative Chest Tube Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Medela AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 1411014891
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Lung Resection
Keywords: Chest tube

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Reg pressure, Active suction (Dig) (Experimental): Regulated pleural pressure with active suction
  Interventions: Other: Reg Pressure; Other: Active Suction (Dig)
- Reg pressure, Passive drainage (Dig) (Experimental): Regulated pleural pressure with passive drainage
  Interventions: Other: Reg Pressure; Other: Passive Drainage (Dig)
- Unreg pressure, Active suction (Trad) (Experimental): Unregulated pleural pressure with active suction
  Interventions: Other: Unreg Pressure; Other: Active Suction (Trad)
- Unreg pressure, Passive drainage (Trad) (Experimental): Unregulated pleural pressure with passive drainage
  Interventions: Other: Unreg Pressure; Other: Passive Drainage (Trad)

INTERVENTIONS:
Other: Reg Pressure — Regulated Suction using the Thopaz+ digital chest drainage device
  Arms: Reg pressure, Active suction (Dig); Reg pressure, Passive drainage (Dig)
Other: Unreg Pressure — Unregulated Suction using a traditional system (multi-chambered system e.g. Pleur-Evac, Atrium-Maquet or similar device as is routine at each institution)
  Arms: Unreg pressure, Active suction (Trad); Unreg pressure, Passive drainage (Trad)
Other: Active Suction (Dig) — Thopaz+ digital chest drainage device set at -20cmH2O at the patient
  Arms: Reg pressure, Active suction (Dig)
Other: Active Suction (Trad) — Pleur-Evac, Atrium-Maquet or similar set at -20cmH2O at the device.
  Arms: Unreg pressure, Active suction (Trad)
Other: Passive Drainage (Dig) — Thopaz+ digital chest drainage device set at -8cmH2O at the patient ("physiologic")
  Arms: Reg pressure, Passive drainage (Dig)
Other: Passive Drainage (Trad) — Pleur-Evac, Atrium-Maquet or similar set by gravity ("water-seal')
  Arms: Unreg pressure, Passive drainage (Trad)

SUMMARY:
A 2 x 2 randomized study testing active versus passive drainage and regulated versus unregulated pleural pressure in patients undergoing anatomic lung resection

DETAILED DESCRIPTION:
This study is a prospective, multi-center randomized clinical trial at 6 sites. Pre-operative evaluation and the decision for surgical intervention will proceed as currently performed at each center. That is, neither inclusion in nor exclusion from this study will affect the plan of care for patients other than the approach to chest tube management, which is determined by randomization among 4 methods that are in common clinical use. Each enrolled patient will be randomized to either regulated pleural pressure using the Thopaz+ digital chest drainage device or unregulated pleural pressure using a traditional system (multi-chambered system e.g. Pleur-Evac, Atrium-Maquet or similar device as is routine at each institution) and also randomized to either active suction (-20 cm H2O) or passive drainage.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to read, understand, and provide written consent
* Age 18-90
* Undergoing a segmentectomy, lobectomy, or bilobectomy (including sleeve resection). Both open and minimally invasive (thoracoscopic or robotic) resections are acceptable

Exclusion Criteria:

* Patients unstable enough to require ICU care for hemodynamic or respiratory problems during the first 7 days postoperatively. Patients admitted to the ICU for other reasons (e.g. bed availability, institutional norm, routine monitoring etc.) should NOT be excluded
* Patients undergoing non-anatomic lung resection only (i.e. wedge resection)
* Patients undergoing anatomic lung resection for bullous disease, lung abscess or bronchiectasis.
* Patients undergoing pneumonectomy or completion pneumonectomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Duration of air leak | up to 7 days
  Duration until there is no clinically significant air leak by standard criteria (no bubbles during coughing with a traditional device and a ≥6 hour period with no spikes >80 ml/min and an air flow ≤30 ml/min during passive drainage or ≤50 ml/min during active suction)

SECONDARY OUTCOMES:
Time till chest tube removal | up to 7 days
  Duration of time till chest tube is removed. Chest tube will be removed when resolution of air leak and fluid drainage <= 400 ml/day

OTHER OUTCOMES:
Duration of hospital stay | up to 7 days
  How long is the total hospital stay
Amount of fluid drained | up to 7 days
  How much fluid is drained while the chest tube is in place

CONTACTS AND LOCATIONS:
Overall Officials: Frank Detterbeck, MD, Principal Investigator — Yale University
Locations (5):
- United States (5):
  - Yale University, New Haven, Connecticut
  - WellStar Health System - Kennestone, Marietta, Georgia
  - Beth Israel Deaconess/ Harvard, Boston, Massachusetts
  - Valley Health System, Paramus, New Jersey
  - St. Luke's Hospital, Bethlehem, Pennsylvania